CLINICAL TRIAL: NCT05991856
Title: Resident Doctor, Master Degree Candidate
Brief Title: Multifaceted Comparison of Ultrasound-guided Ablation and Laparoscopic Adrenalectomy for Aldosterone-producing Adenoma
Status: Recruiting | Type: Observational
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xubin Yang, Dr., Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: HuanXu
Record Dates: First submitted 2023-07-23; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Aldosterone-producing Adenoma; Radiofrequency Ablation
Keywords: aldosterone-producing adenoma; radiofrequency ablation; laparoscopic adrenalectomy
MeSH Terms: conditions — Adrenocortical Adenoma | interventions — Radiofrequency Ablation; Antihypertensive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- radiofrequency ablation: Patients with aldosterone-producing adenoma undergoing ultrasound-guided radiofrequency ablation
  Interventions: Procedure: radiofrequency ablation; Drug: Hypotensive Drugs
- laparoscopic adrenalectomy: Patients with aldosterone-producing adenoma undergoing laparoscopic adrenalectomy
  Interventions: Procedure: laparoscopic adrenalectomy; Drug: Hypotensive Drugs

INTERVENTIONS:
Procedure: radiofrequency ablation — The subjects is placed in a prone or lateral position under local anesthesia, and the electrodes are placed in the adrenal nodules under ultrasound guidance. A rapidly alternating radiofrequency current (300-500khz) generated around the electrode propagates through the adrenal nodules, causing resistance heating (Joule effect) and inducing cell death through coagulation necrosis. The choice of ablation time and frequency depends on the size, shape and location of the nodules within the adrenal gland.
  Other Names: RFA
  Groups: radiofrequency ablation
Procedure: laparoscopic adrenalectomy — The subjects was placed in a lateral position under general anesthesia. Using harmonic scalpel carefully separates the adrenal vessels and lates them. The adipose tissue around the adrenal gland is dissected carefully, the surrounding tissue is bluntly separated, and the adrenal gland is fully exposed and dissected. After adrenalectomy was completed, hemostasis was rechecked and specimens were removed.
  Other Names: LA
  Groups: laparoscopic adrenalectomy
Drug: Hypotensive Drugs — All subjects in the study selected appropriate antihypertensive drugs based on factors such as blood pressure level.
  Other Names: HD

SUMMARY:
The purpose of this study is to retrospectively and prospectively analyze the efficacy and safety of ultrasound-guided radiofrequency ablation and laparoscopic adrenalectomy in the treatment of aldosterone-producing adenoma (APA). It is planned to retrospectively collect 30 patients with adrenal radiofrequency ablation for APA and 15 patients with age - and sex-matched laparoscopic adrenalectomy for APA in our hospital from January 2020 to June 2024, and continue to follow up for 3 years.

DETAILED DESCRIPTION:
Primary aldosteronism is the most common cause of secondary hypertension, and aldosterone-producing adenoma (APA) is a benign adrenal tumor, accounting for about 35% of primary aldosteronism. According to clinical guidelines, laparoscopic adrenalectomy is the preferred treatment for unilateral APA. Recently, radiofrequency ablation, as a new technique, has been applied to the treatment of APA. However, there are few relevant studies, the sample size is generally small, and basically belong to retrospective studies, lacking the comparison of long-term postoperative effects. Our hospital is the first to carry out ultrasound-guided radiofrequency ablation of APA in Guangdong, China, with satisfactory results. The purpose of this study is to retrospectively and prospectively analyze the efficacy and safety of ultrasound guided radiofrequency elimination and laparoscopic adrenalectomy in the treatment of APA. It is planned to retrospectively collect 30 patients with adrenal radiofrequency ablation for APA and 15 patients with age - and sex-matched laparoscopic adrenalectomy for APA in our hospital from January 2020 to June 2024, and continue to follow up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. APA was confirmed with unilateral lesions;
2. Benign tumor without adrenal metastasis and endovascular tumor embolus;
3. Receive ultrasound-guided adrenal RFA treatment or laparoscopic resection, and sign the informed consent for surgery;
4. Age ≥ 18;
5. Age ≥ 40 years old should meet the following criteria: blood potassium ≤3.5mmol/L; PAC≥20ng/dL; PRC≤5μIU/mL; A unilateral adrenal nodule of 10mm or more was completely normal on the opposite side.

Exclusion Criteria:

1. Bilateral adrenal diseases;
2. Multiple adrenal tumors;
3. Other adrenal diseases, such as adrenal hyperplasia, Cushing's syndrome, pheochromocytoma, etc.;
4. Imaging suggests that the tumor may be difficult to reach;
5. Imaging showed potential malignant adrenal tumor;
6. Pregnant and/or planning a pregnancy;
7. Refusing to participate in follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2020 to January 2024, patients with APA were treated with adrenal RFA in our hospital
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Within 3 years
  Effect of radiofrequency ablation and laparoscopic adrenalectomy on blood pressure levels in aldosterone-producing adenoma patients, including systolic and diastolic blood pressure(in millimeters of mercury, mmHg).
Serum potassium | Within 3 years
  Effect of radiofrequency ablation and laparoscopic adrenalectomy on serum potassium (mmol/L) levels in aldosterone-producing adenoma patient.
Aldosterone | Within 3 years
  The effects of radiofrequency ablation and laparoscopic adrenalectomy on aldosterone levels(ng/dl) in aldosterone-producing adenoma patients.
ARR | Within 3 years
  The effects of radiofrequency ablation and laparoscopic adrenalectomy on ARR (plasma aldosterone to renin activity ratio) in aldosterone-producing adenoma patients.
Complications | Within 3 years
  Intraoperative or postoperative complications of both types of surgery, including hypertensive crises, bleeding, and pancreatitis.
PASO | Within 3 years
  PASO(the Primary Aldosteronism Surgical Outcome) criteria were used to standardize the evaluation of outcomes of radiofrequency ablation and laparoscopic adrenalectomy, divided into clinical and biochemical outcomes, and the outcome grades were defined in terms of complete success, partial success, and unsuccessful.

SECONDARY OUTCOMES:
Operation cost | Within 3 years
  Comparison of the operation costs of radiofrequency ablation and laparoscopic adrenalectomy.
Length of hospital stays | Within 3 years
  Comparison of the hospital stays of radiofrequency ablation and laparoscopic adrenalectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Mengyin Cai, Dr, Study Chair — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Background] Brown JM, Siddiqui M, Calhoun DA, Carey RM, Hopkins PN, Williams GH, Vaidya A. The Unrecognized Prevalence of Primary Aldosteronism: A Cross-sectional Study. Ann Intern Med. 2020 Jul 7;173(1):10-20. doi: 10.7326/M20-0065. Epub 2020 May 26. PMID 32449886
- [Background] Williams TA, Lenders JWM, Mulatero P, Burrello J, Rottenkolber M, Adolf C, Satoh F, Amar L, Quinkler M, Deinum J, Beuschlein F, Kitamoto KK, Pham U, Morimoto R, Umakoshi H, Prejbisz A, Kocjan T, Naruse M, Stowasser M, Nishikawa T, Young WF Jr, Gomez-Sanchez CE, Funder JW, Reincke M; Primary Aldosteronism Surgery Outcome (PASO) investigators. Outcomes after adrenalectomy for unilateral primary aldosteronism: an international consensus on outcome measures and analysis of remission rates in an international cohort. Lancet Diabetes Endocrinol. 2017 Sep;5(9):689-699. doi: 10.1016/S2213-8587(17)30135-3. Epub 2017 May 30. PMID 28576687
- [Background] Yang MH, Tyan YS, Huang YH, Wang SC, Chen SL. Comparison of radiofrequency ablation versus laparoscopic adrenalectomy for benign aldosterone-producing adenoma. Radiol Med. 2016 Oct;121(10):811-9. doi: 10.1007/s11547-016-0662-1. Epub 2016 Jun 14. PMID 27300650